CLINICAL TRIAL: NCT00353860
Title: Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation Followed by T Cell Add-Back for Hematological Malignancies - Role of Preparative Regimen and T Cell Dose in Graft Rejection and GVHD
Brief Title: Stem Cell Transplantation and T-Cell Add-Back to Treat Bone Marrow Malignances
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020111; 02-H-0111
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-11-21

CONDITIONS: Immunosuppression; Leukemia
Keywords: Leukemia; Transplant - Mortality; Immunosuppression; Radiation; Cure; Peripheral Blood Stem Cells; Graft-Versus Leukemia/Myeloma; Graft-Versus-Host Disease; Cyclosporine; Fludarabine
MeSH Terms: conditions — Leukemia; Neoplasms, Plasma Cell; Graft vs Host Disease

INTERVENTIONS:
Device: SOLEX 300i Stem Cell Selection

SUMMARY:
This study will evaluate the safety and effectiveness of stem cell transplantation in which the donor s T cells (a type of lymphocyte, or white blood cell) have been removed and then added back. Certain patients with bone marrow malignancies undergo transplantation of donated stem cells (cells produced by the bone marrow that mature into the different blood components white cells, red cells and platelets) to generate new and normally functioning bone marrow. However, T-cells from the donor may see the patient s cells as foreign and mount an immune response to reject them, causing what is called graft-versus-host-disease (GVHD). Therefore, in this study, T-cells are removed from the donor cells to prevent this complication. Nevertheless, there are disadvantages of removing the T-cells, since they are important in fighting viral infections as well as any remaining malignant cells. The attack against the malignant cells is called a graft-versus-leukemia effect. Therefore, donor T cells are given to the patient (added back) later (45 and 100 days after the transplant) when they can provide needed immunity with less risk of causing GVHD.

Patients between 10 and 55 years of age with chronic myelogenous leukemia, acute lymphoblastic leukemia, acute myelogenous leukemia, a myelodysplastic syndrome, myeloproliferative disorders, or chronic lymphocytic leukemia may be eligible for this study. Prospective participants and their donors are screened with a medical history and physical examination, blood tests (including a test to match for genetic compatibility), breathing tests, chest and sinus X-rays, and tests of heart function. They also undergo a bone marrow biopsy and aspiration. For this procedure, done under local anesthetic, about a tablespoon of bone marrow is withdrawn through a needle inserted into the hipbone.

Participants may undergo apheresis to collect lymphocytes for research studies. This procedure involves collecting blood through a needle in the arm, similar to donating a unit of blood. The lymphocytes are then separated and removed by a cell separator machine, and the rest of the blood is returned through a needle in the other arm.

Before treatment begins, patients have a central venous catheter (flexible plastic tube) placed in a vein. This line remains in place during the stem cell transfusion and recovery period for drawing and transfusing blood, giving medications, and infusing the donated cells. Preparation for the transfusion includes irradiation and chemotherapy. Patients undergo total body irradiation in 8 doses given in two 30-minute sessions a day for 4 days. Four days before the transfusion, they begin taking cyclophosphamide, and 9days before the procedure they start fludarabine. These are anti-cancer drugs that kill the cancer cells and prevent rejection of the donated cells. While the patient is receiving chemotherapy, the donor receives daily injections for 6 days of G-CSF, a drug that moves stem cells from the bone marrow into the blood stream. On days 1 and 2 after chemotherapy is completed, the stem cells are infused into the patient through the central line.

Patients usually stay in the hospital about 20 to 30 days after the transplant to recover from treatment side effects, which may include fever, nausea, diarrhea and mouth pain, and receive blood transfusions, if needed. Treatment with cyclosporine, a drug that helps prevents both rejection of donated cells and GVHD, is started on day 44 one day before the first T-cell add-back. Patients return to the clinic for follow-up with various tests, treatments and examinations as required, with a minimum of visits at least once or twice a week for 2 to 4 months after the transplant; then at 4, 6, 9, and 12 months, and then yearly for at least 3 years.

DETAILED DESCRIPTION:
Bone marrow stem cell transplant studies carried out by the NHLBI BMT Unit have focused on approaches to optimize the stem cell and lymphocyte dose in order to improve transplant survival and increase the graft-vs.-leukemia effect. The aim is to create the transplant conditions that permit rapid donor immune recovery without causing graft-versus-host disease (GVHD) by using no post-transplant immunosuppression in conjunction with a transplant depleted of T cells to a fixed low dose, below the threshold known to be associated with GVHD. A primary objective of the protocol is therefore to test whether the low dose of T cells chosen minimizes the risk and severity of GVHD.

We have found that the outcome from transplant is improved by using high stem cell doses, and in successive protocols we have achieved progressive improvement in transplant-related mortality from 35% in the first protocol in 1993 to 22% for the latest study. In the last study, in this series, we used the Nexell Isolex 300i system to obtain high CD34+ doses depleted of lymphocytes to a fixed CD3+ T cell dose of 5 x 10(4)/kg. The use of the cell separator and the monoclonal antibodies is covered by IDE 8139. The study focused on the role of cyclosporine in preventing GVHD after T cell depletion. We found that CSA appears to protect against both GVHD and graft failure, with a higher incidence of both complications occurring in patients not receiving CSA.

To address the results and shortcomings of the previous protocol, while continuing to avoid immunosuppression post-transplant, we will now test two hypotheses: (1) GVHD incidence and severity can be reduced by transfusing a T cell dose of 2 x 10(4)/CD3 cell/kg. (2) Graft rejection can be prevented by increasing the immunosuppressive intensity of the pre-transplant preparative regimen using fludarabine and cyclophosphamide and a reduced dose of total body irradiation (12 Gy instead of 13.6 Gy). We will use the same in vitro cell separation system namely the Isolex 300i and monoclonal antibodies provided by CTEP (anti CD 6, anti CD2, anti CD7). This is covered by a continuing IND for the selection of CD34+ and CD3+ cells for T cell depleted peripheral blood stem cell transplantation.

ELIGIBILITY:
* INCLUSION CRITERIA - PATIENT:

Ages 10-55 years inclusive (but less than 56).

Chronic myelogenous leukemia in chronic phase

A) Patients not treated with STI 571 under the age of 41 (subject to regular DSMB review);

B) Age 10-55 in chronic phase who have failed treatment with STI-571;

C) Age 10-55 in accelerated phase or blast transformation.

Acute lymphoblastic leukemia, any of these categories: Adults (greater than 18 years) in first remission with high-risk features (presenting leukocyte count greater than 100,000/cu mm, karyotypes t9; 22, t4, t19, t11, biphenotypic leukemia). All second or subsequent remissions, primary induction failure, partially responding or untreated relapse.

Acute myelogenous leukemia (AML): AML in first remission except AML with good risk karyotypes: AML M3 (t15; 17), AML M4Eo (inv 16), AML t (8; 21). All AML in second or subsequent remission, primary induction failure and resistant relapse.

Myelodysplastic syndromes, any of these categories: refractory anemia with transfusion dependence, refractory anemia with excess of blasts, transformation to acute leukemia, chronic myelomonocytic leukemia.

Myeloproliferative disorders (myelofibrosis, polycythemia vera, essential thrombocythemia) in transformation to acute leukemia.

Chronic lymphocytic leukemia refractory to fludarabine treatment and with bulky progressive disease or with thrombocytopenia (less than or equal to 100,000/microliters) or anemia (less than or equal to 10 g/dl) not due to recent chemotherapy.

No major organ dysfunction precluding transplantation.

DLCO greater than or equal to 60% predicted.

Left ventricular ejection fraction: greater than or equal to 40% predicted.

ECOG performance status of 0 or 1.

For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian. Informed oral consent from minors: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

Negative pregnancy test for women of childbearing age.

INCLUSION CRITERIA - DONORS:

HLA 6/6 identical family donor.

Weight greater than or equal to 18 kg.

Age less than or equal to 80 years old.

Fit to receive G-CSF and give peripheral blood stem cells (normal blood count, normotensive, no history of stroke).

For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian and informed assent: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

EXCLUSION CRITERIA - RECIPIENT:

Patient pregnant.

Age less than 10 years and 56 years or more.

Patients with CML in chronic phase who are 41 years or over in whom STI 571 is the treatment of choice.

ECOG performance status of 2 or more.

Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible.

Major anticipated illness or organ failure incompatible with survival from BMT.

DLCO less than 60% predicted.

Left ventricular ejection fraction: less than 40% predicted.

Serum creatinine greater than 3 mg/dl.

Serum bilirubin greater than 4 mg/dl.

Transaminases greater than 3x upper limit of normal.

HIV positive.

History of other malignancies except basal cell or squamous carcinoma of the skin, positive PAP smear and subsequent negative follow up.

Individuals with diseases listed in the inclusion criteria but where debility or age makes the risk of intensive myeloablative therapy unacceptable. This includes patients who have received busulfan treatment for more than 6 months continuously. These patients will be considered for non-myeloablative allogeneic transplantation protocols.

EXCLUSION CRITERIA - DONOR

Pregnant or lactating.

Donor unfit to receive G-CSF and undergo apheresis. (uncontrolled hypertension, history of congestive heart failure, or unstable angina, thrombocytopenia).

HIV positive. Donors who are positive for HBV, HCV or HTLV-1 may be used if the risk-benefit ratio is considered acceptable by the patient and investigator.

Weight less than 18 kg.

Age greater than 80 years.

Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the BMT treatment unlikely, and making informed consent impossible.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-01-23; Primary Completion 2007-11-29 (Actual); Study Completion 2007-11-29 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with clinically significant acute GHVD (Grade II or higher) following the T depleted PBPC transplant. | Before day 45.

CONTACTS AND LOCATIONS:
Overall Officials: A. John Barrett, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Couriel D, Canosa J, Engler H, Collins A, Dunbar C, Barrett AJ. Early reactivation of cytomegalovirus and high risk of interstitial pneumonitis following T-depleted BMT for adults with hematological malignancies. Bone Marrow Transplant. 1996 Aug;18(2):347-53. PMID 8864445
- [Background] Mavroudis D, Read E, Cottler-Fox M, Couriel D, Molldrem J, Carter C, Yu M, Dunbar C, Barrett J. CD34+ cell dose predicts survival, posttransplant morbidity, and rate of hematologic recovery after allogeneic marrow transplants for hematologic malignancies. Blood. 1996 Oct 15;88(8):3223-9. PMID 8874224
- [Background] Mavroudis DA, Read EJ, Molldrem J, Raptis A, Plante M, Carter CS, Phang S, Dunbar CE, Barrett AJ. T cell-depleted granulocyte colony-stimulating factor (G-CSF) modified allogenic bone marrow transplantation for hematological malignancy improves graft CD34+ cell content but is associated with delayed pancytopenia. Bone Marrow Transplant. 1998 Mar;21(5):431-40. doi: 10.1038/sj.bmt.1701120. PMID 9535034
- [Derived] McIver ZA, Yin F, Hughes T, Battiwalla M, Ito S, Koklanaris E, Haggerty J, Hensel NF, Barrett AJ. Second hematopoietic SCT for leukemia relapsing after myeloablative T cell-depleted transplants does not prolong survival. Bone Marrow Transplant. 2013 Sep;48(9):1192-7. doi: 10.1038/bmt.2013.39. Epub 2013 Mar 25. PMID 23524640
- [Derived] McIver Z, Melenhorst JJ, Wu C, Grim A, Ito S, Cho I, Hensel N, Battiwalla M, Barrett AJ. Donor lymphocyte count and thymic activity predict lymphocyte recovery and outcomes after matched-sibling hematopoietic stem cell transplant. Haematologica. 2013 Mar;98(3):346-52. doi: 10.3324/haematol.2012.072991. Epub 2012 Oct 12. PMID 23065508